CLINICAL TRIAL: NCT05819983
Title: Comparison of Effectiveness Between Three Dosages of Oral Ivermectin, Two Dosages of Oral Ivermectin, and Two Applications of Topical Permethrin In Scabies Patients
Brief Title: Ivermectin/ Permethrin for Scabies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DV202303.01
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Scabies
MeSH Terms: conditions — Scabies | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral ivermectin 3 dosages and placebo (Active Comparator): Twenty patients will be administered randomly oral ivermectin 200µg/kg BW on days 1, 2, and 8 and also placebo cream on days 1 and 8
  Placebo cream: Cream base
  Interventions: Drug: Ivermectin Tablets
- Oral ivermectin 2 dosages and placebo (Active Comparator): Twenty patients will be administered randomly oral ivermectin 200µg/kg BW on days 1 and 8 and also oral placebo on day 2, placebo cream on days 1 and 8
  Placebo cream: Cream base
  Interventions: Drug: Ivermectin Tablets
- Permethrin 5% cream 2 applications and placebo (Active Comparator): Twenty patients will be administered randomly permethrin 5% cream on days 1 and 8 and also oral placebo on days 1, 2, and 8
  Placebo: vitamin B complex
  Interventions: Drug: Permethrin Cream

INTERVENTIONS:
Drug: Ivermectin Tablets — Ivermectin 200µg/kg BW
  Arms: Oral ivermectin 2 dosages and placebo; Oral ivermectin 3 dosages and placebo
Drug: Permethrin Cream — Permethrin cream 5%
  Arms: Permethrin 5% cream 2 applications and placebo

SUMMARY:
Scabies is a skin disease characterized by intense itching that worsens at night. It is very contagious, still has a high occurrence rate, and impacts patient quality of life. The use of scabicide followed by a clean and healthy lifestyle is the principle of scabies therapy. The primary treatment option for scabies is permethrin 5% cream. Ivermectin is an alternate treatment for scabies.

DETAILED DESCRIPTION:
Permethrin acts by disrupting the sodium channel current, resulting in delayed repolarization, paralysis, and death of the parasite. Sodium channels are ubiquitous and therefore permethrin acts at all stages of the life cycle of the parasite. Permethrin 5% cream is applied overnight once a week for two weeks to the entire body. This drug has a number of negative side effects, such as being expensive, uncomfortable, less applicable, and in some cases resistant to permethrin. Ivermectin is an alternate treatment for scabies and should be administered twice, one week apart. Ivermectin acts by binding selectively and with high affinity to glutamate-gated chloride ion channels, which are present in invertebrate nerve and muscle cells, resulting in paralysis and death of the parasite. Two doses of ivermectin one week apart are recommended for scabies treatment. Due to its specific site of action, ivermectin may not be effective against the younger stages of the parasite inside the egg because the nervous system has not yet developed. This drug is safe, more affordable, more practical to use, and has minimal side effects. The disadvantage of ivermectin is it does not kill all the stages of S. scabiei, necessitating multiple doses. According to several earlier research, topical permethrin is just as effective as oral ivermectin at one or two doses.

There hasn't been any research on how well three doses of oral ivermectin treat scabies. As a result of no data, our trial is looking forward to answering the comparison of the effectiveness between three dosages of oral ivermectin, two dosages of oral ivermectin, and two applications of topical permethrin in scabies patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 6 years or above
* Body weight 15kg or above
* Clinical establishment of diagnosed scabies

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Scabies with secondary infection
* Scabies with eczematization
* History of receiving scabies treatment in the last four weeks
* History of drug hypersensitivity

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
The severity of scabetic lesions | 5 weeks
  Determined by counting the number of lesions and graded as:
  0 = Free of lesions (no scabies) 10 or fewer lesions = Mild 11-49 lesions= Moderate 50 or more lesions= Severe
The severity of pruritus | 5 weeks
  Evaluated by the patients graded on a scale 0-10 (using VAS score):
  0= No pruritus 1-3= Mild 4-6= Moderate 7-10= Severe

SECONDARY OUTCOMES:
Clinical improvement | 4 weeks
  Defined as a reduction in both the number of lesions and symptoms and graded as:
  Mild= Less than 50% reduction in the number of lesions and pruritus Moderate= More than or equal to 50% reduction in the number of lesions and pruritus Good= Complete clearance of the lesion and pruritus
Side effects | 4 weeks
  Evaluated the side effects after using oral ivermectin or permethrin 5% cream.

CONTACTS AND LOCATIONS:
Overall Officials: Hendra Gunawan,, M.D., PhD, Principal Investigator — Faculty of Medicine Universitas Padjadjaran Bandung
Locations (1):
- Ciumbuleuit Public Health Centre, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided